CLINICAL TRIAL: NCT01636596
Title: Evaluating the Efficacy of Controlled Pulsatile Intravenous Insulin on Cognition and Amyloid Burden in Patients With Alzheimer's Disease- A Pilot Study
Brief Title: Efficacy of Pulsatile IV Insulin on Cognition and Amyloid Burden in Patients With Alzheimer's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Acuity Center (Unknown)
Responsible Party: Principal Investigator, James C. Patterson, II, MD. Ph, Professor Psychiatry, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12-166
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Insulin; Pulsatile
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Insulin Resistance | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Insulin LISPRO — Insulin is delivered in a pulsatile fashion. One treatment is approximately 10-15 units of insulin (exact dose based on weight) split into ten pulses delivered over one hour. Three treatments will be administered per session with one session per week for six month duration.
  Other Names: Humalog

SUMMARY:
The objectives of this project are to examine amyloid burden and cognition in a group of subjects diagnosed with Alzheimer's Disease (AD) or Mild Cognitive Impairment (MCI) before and after a six month course of insulin delivered weekly in a controlled pulsatile intravenous fashion in a clinical setting. The investigators central hypothesis is straightforward: The investigators predict that controlled pulsed IV infusion of insulin will improve cognition in patients with AD, and that this improvement will be correlated with a decrease in amyloid burden in these patients.

DETAILED DESCRIPTION:
Visit 1: Consent/Assent will be obtained before any study related procedures are performed. Once consent is obtained subjects will be assessed to determine eligibility based on study inclusion/exclusion criteria. A history and physical with possible neurological examination will be conducted. Cognitive impairment will be assessed by having the subject complete the Folstein Mini-Mental State Exam (MMSE).

Qualifying subjects who wish to participate in the study will be scheduled to return for a study orientation visit. Subjects are required to have a study partner. Subjects will be given a copy of the study partner informed consent form (ICF) to take home with them. A potential study partner(s) must attend the orientation visit with the subject.

Visit 2: Study Orientation: ICF will be obtained from subject study partner(s). Subjects and their study partner(s) will be given information about what is required for the study. They will be given the patient logs that are to be kept at home between sessions and discussed with study staff at the following session. Subjects and study partners will be trained to become proficient in checking their blood sugar with one of the common blood glucose meters as well as how to use a supply of glucose which can cover any potential hypoglycemic reaction. Subjects and/or their study partners will be oriented to the location where the controlled pulsatile IV insulin infusion therapy will be performed. They will be instructed on where to park and where to go when they arrive.

Visit 3: Pre-Therapy Amyloid PET scan

Visits 4 - 28: Insulin Therapy Visits: Subjects will complete 25 insulin therapy sessions which will occur on a weekly basis, over 6 months. Prior to insulin treatment the following assessments will be completed: MMSE, CDT, QOLS, and CGI. Also prior to insulin therapy, as well as between insulin therapy treatments, basal O2 and C O2 measurements will be obtained.

Pre labs will be collected at visit 4, mid labs at visit 16, and post labs at visit 28.

Visit 29: Post-therapy Amyloid PET Scan

Visit 30: The final study visit will be conducted in the Psychopharmacology Research Clinic within one month of the subject completing the last insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 and 95 years of age
* Have a clinical diagnosis of Mild Cognitive Impairment or Alzheimer's Disease
* Have a Folstein Mini-Mental State Exam (MMSE) score of 15 or greater
* Be physically able to take part in the study
* Females will not be of child-bearing potential (one year postmenopausal, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)
* Be able to give informed consent for study procedures; if incapable of giving informed consent, the subject's designated decision maker may consent on their behalf but the subject must still be able to confirm assent
* Have a "study partner" willing to accompany them to all study visits

Exclusion Criteria:

* Have a major or unstable medical illness such that, in the PI's clinical judgment, will prohibit or interfere with involvement in this research protocol, including diabetes
* Have current substance or alcohol dependence, or abuse within the last eight weeks
* Have the ApoE4 homozygous genotype

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
cerebral glucose metabolism | 25 weeks
  Cerebral glucose metabolism will be measured using pre and post FDG PET Scans.
cognition | 30 weeks
  Changes in cognition will be measured before therapy, on a weekly basis during therapy, and after therapy using the Folstein Mini-Mental State Exam (MMSE) and the Clock Drawing Test (CDT).

SECONDARY OUTCOMES:
general clinical improvement | 30 weeks
  Changes in general clinical improvement will be measured before therapy, on a weekly basis during therapy, and after therapy using the Clinical Global Impression (CGI) and the Quality of Life Scale (QOLS).
basal metabolism | 30 weeks
  Changes in basal metabolism will be measured before therapy, during weekly treatment sessions, and after therapy using measured O2 and CO2 levels.

CONTACTS AND LOCATIONS:
Overall Officials: James C Patterson, MD PhD, Principal Investigator — LSUHSC Shreveport
Locations (1):
- LSUHSC Shrevport Psychopharmacology Research Clinic, Shreveport, Louisiana, United States